CLINICAL TRIAL: NCT03700086
Title: Efficacy of a Disposable Negative Wound Pressure Device in Reducing the Incidence of Non-organ Space Surgical Site Infection After Clean-contaminated Pancreatic Resections: a Randomized Controlled Trial
Brief Title: Efficacy of NPWT in Reducing the Incidence of Wound Infection After Pancreatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Smith & Nephew Wound Management Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PICO (1215CESC)
Record Dates: First submitted 2018-05-15; First posted 2018-10-09 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-03

CONDITIONS: Surgical Site Infection
Keywords: negative pressure wound therapy; wound infection; pancreaticoduodenectomy; total pancreatectomy; surgical palliation of pancreatic cancer
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Negative wound pressure device (PICO) (Experimental): The disposable negative wound pressure device (PICO) will be used to cover the midline incision. The dressing is changed on POD3 and removed on POD7. Data are collected on POD3, POD7 and POD30.
  Interventions: Device: Disposable negative wound pressure device (PICO)
- Standard sterile dressing (Active Comparator): The OPsite post-op visible standard sterile dressing will be used to cover the midline incision. Dressing is changed q48h. Data are collected on POD3, POD7 and POD30.
  Interventions: Device: OPsite post-op visible standard sterile dressing

INTERVENTIONS:
Device: Disposable negative wound pressure device (PICO) — Application of a disposable negative wound pressure device for surgical site infection prevention.
  Arms: Negative wound pressure device (PICO)
Device: OPsite post-op visible standard sterile dressing — Application of a standard sterile wound dressing.
  Arms: Standard sterile dressing

SUMMARY:
A disposable negative wound pressure device will be compared to standard sterile wound dressing in reducing the rate of wound infection after clean-contaminated surgical procedures on biliary tract and pancreas in patients at high risk for wound infection.

DETAILED DESCRIPTION:
The use of specific protocols for antisepsis, sterilization and infections' prophylaxis is widely diffused, but, however, surgical site infection rate is still high. Wound infection is often considered as a minor morbidity if compared with other complications, but it is able to considerably increase the length of hospital stay, health care and assistance related costs affecting patients' quality of life. The Center for Disease Control and Prevention (CDC) has published specific guidelines for surgical site infection (SSI) prevention that includes hairs removal, intravenous antibiotics on the basis of the type of procedure planned for that patient, skin antisepsis, surgical team antisepsis, sterility, blood glucose levels control, body temperature control and optimal perfusion of all tissues. At the end of the surgical procedure, surgical incision is covered with a sterile dressing that usually is changed after 24/48 hours. Clean-contaminated procedures like pancreaticoduodenectomy (PD), total pancreatectomy (TP) and palliative procedures like gastric by-pass and hepaticojejunostomy GEA/HJ) are considered at high complexity with a high incidence of SSI, especially dealing with patients at high surgical risk. Since from the introduction of negative wound pressure therapy in 1997, these devices have been used only for the treatment of acute and chronic wounds with loss of tissue, but recently have also been proposed in the setting of SSI prevention. Negative wound pressure systems have higher costs, the use in the outpatients setting may be complex consequently the use in the setting of SSI prevention could not result cost-effective.

The rationale for the use of negative pressure therapy in the prevention of SSI relies in the complete clearance of dead-space under the incision, fluids and blood removal with consequent reduction of fluids infections, edema reduction, blood flow improvement and tissue oxygenation. Similar results can be obtained through a less expensive, disposable, canisterless, negative pressure wound therapy device (Pico®, Smith&Nephew). This system is cheaper, is portable, and can produce a continue vacuum with a nominal pressure of -80mmHg being able to achieve a rapid discharge at home with less frequent medications, improved comfort and aesthetic result.

The following study is designed to assess the effect of a disposable, canisterless, negative pressure wound therapy device in the reduction of SSI in high risk patients if compared with a sterile standard dressing after major pancreatic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Informed consent
* HPB clean-contaminated procedures (PD, TP and GEA/HJ)
* Median laparotomy
* Compliance with a follow-up protocol
* High risk for SSI (at least one of the following):

  * Body Mass Index > 30kg/m2
  * Diabetes mellitus type I or II
  * Use of steroids
  * Neoadjuvant therapy
  * ASA ≥ 3
  * Charlson Comorbidity Index 1
  * Time of surgery > 360'
  * Estimated blood loss > 1L

Exclusion Criteria:

* Previous open surgery of the abdomen
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (non-organ space) | 30 days from index surgery
  Superficial + deep surgical site infection as defined by CDC

SECONDARY OUTCOMES:
Rate of discontinuation of negative wound pressure therapy | 7 days from index surgery
  Discontinuation of therapy due to patient choice
Incidence of seromas | 30 days from index surgery
  As defined by CDC
Incidence of hematomas | 30 days from index surgery
  As defined by CDC
Incidence of major morbidities | 30 days from index surgery
  Incidence of pancreatic fistula, hemorrhage, delayed gastric emptying, Clavien -Dindo morbidity
Stony Brook Scar Evaluation Scale Score | 30 days after index surgery
  The Stony Brook Evaluation Scale evaluate the aesthetic result of an incision. Score ranges from 0 (worst aesthetic result) to 5 (best aesthetic result)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Landoni, MD, Principal Investigator — AOVR Veneto
Locations (1):
- Ospedale Policlinico GB Rossi, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fiorio M, Marvaso A, Vigano F, Marchetti F. Incidence of surgical site infections in general surgery in Italy. Infection. 2006 Dec;34(6):310-4. doi: 10.1007/s15010-006-6632-0. PMID 17180584
- [Result] Allegranzi B, Bagheri Nejad S, Combescure C, Graafmans W, Attar H, Donaldson L, Pittet D. Burden of endemic health-care-associated infection in developing countries: systematic review and meta-analysis. Lancet. 2011 Jan 15;377(9761):228-41. doi: 10.1016/S0140-6736(10)61458-4. Epub 2010 Dec 9. PMID 21146207
- [Result] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Result] Ceppa EP, Pitt HA, House MG, Kilbane EM, Nakeeb A, Schmidt CM, Zyromski NJ, Lillemoe KD. Reducing surgical site infections in hepatopancreatobiliary surgery. HPB (Oxford). 2013 May;15(5):384-91. doi: 10.1111/j.1477-2574.2012.00604.x. Epub 2012 Nov 5. PMID 23557410
- [Result] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Result] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Result] Masden D, Goldstein J, Endara M, Xu K, Steinberg J, Attinger C. Negative pressure wound therapy for at-risk surgical closures in patients with multiple comorbidities: a prospective randomized controlled study. Ann Surg. 2012 Jun;255(6):1043-7. doi: 10.1097/SLA.0b013e3182501bae. PMID 22549748
- [Result] Vargo D. Negative pressure wound therapy in the prevention of wound infection in high risk abdominal wound closures. Am J Surg. 2012 Dec;204(6):1021-3; discussion 1023-4. doi: 10.1016/j.amjsurg.2012.10.004. PMID 23231938
- [Result] Blackham AU, Farrah JP, McCoy TP, Schmidt BS, Shen P. Prevention of surgical site infections in high-risk patients with laparotomy incisions using negative-pressure therapy. Am J Surg. 2013 Jun;205(6):647-54. doi: 10.1016/j.amjsurg.2012.06.007. Epub 2013 Jan 30. PMID 23375758
- [Result] Bonds AM, Novick TK, Dietert JB, Araghizadeh FY, Olson CH. Incisional negative pressure wound therapy significantly reduces surgical site infection in open colorectal surgery. Dis Colon Rectum. 2013 Dec;56(12):1403-8. doi: 10.1097/DCR.0b013e3182a39959. PMID 24201395
- [Result] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014
- [Result] Webster J, Scuffham P, Sherriff KL, Stankiewicz M, Chaboyer WP. Negative pressure wound therapy for skin grafts and surgical wounds healing by primary intention. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD009261. doi: 10.1002/14651858.CD009261.pub2. PMID 22513974
- [Result] Malmsjo M, Huddleston E, Martin R. Biological effects of a disposable, canisterless negative pressure wound therapy system. Eplasty. 2014 Apr 2;14:e15. eCollection 2014. PMID 24741386
- [Result] Fong ZV, McMillan MT, Marchegiani G, Sahora K, Malleo G, De Pastena M, Loehrer AP, Lee GC, Ferrone CR, Chang DC, Hutter MM, Drebin JA, Bassi C, Lillemoe KD, Vollmer CM, Fernandez-Del Castillo C. Discordance Between Perioperative Antibiotic Prophylaxis and Wound Infection Cultures in Patients Undergoing Pancreaticoduodenectomy. JAMA Surg. 2016 May 1;151(5):432-9. doi: 10.1001/jamasurg.2015.4510. PMID 26720272
- [Result] Payne C, Edwards D. Application of the Single Use Negative Pressure Wound Therapy Device (PICO) on a Heterogeneous Group of Surgical and Traumatic Wounds. Eplasty. 2014 Apr 28;14:e20. eCollection 2014. PMID 24917894
- [Result] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Am J Infect Control. 1992 Oct;20(5):271-4. doi: 10.1016/s0196-6553(05)80201-9. No abstract available. PMID 1332552
- [Result] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Result] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Result] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Result] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Result] Pellino G, Sciaudone G, Candilio G, Campitiello F, Selvaggi F, Canonico S. Effects of a new pocket device for negative pressure wound therapy on surgical wounds of patients affected with Crohn's disease: a pilot trial. Surg Innov. 2014 Apr;21(2):204-12. doi: 10.1177/1553350613496906. Epub 2013 Jul 24. PMID 23883481